CLINICAL TRIAL: NCT04551794
Title: iCBT for Depression: A Randomized Controlled Trial Comparing Different Levels of Guidance
Brief Title: Different Levels of Guidance in iCBT for Depression (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Selfapy
Record Dates: First submitted 2020-08-29; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Depressive Symptoms; Quality of Life; Self Esteem
Keywords: Depressive symptoms, iCBT, guidance, peer-support, RCT
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled study with three conditions: Condition 1: Online intervention with therapeutic guidance (telephone contacts). Condition 2: Online intervention with additional peer support (online forum). Condition 3: Wait-list control group (access to the online intervention after completion of the post-assessment).
  Two assessments-points, the intervention period (pre-post) is three months. At both assessments psychopathological data are obtained via the Internet survey Enterprise Feedback Suite survey by QuestBack Unipark®.
Masking Description: Masking was not necessary as the participants were automatically randomized within the baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online self-help program with additional peer support (Experimental): The intervention group receives the login data for the online program directly following the baseline assessment. The program consists of 9 modules with many interactional exercises. Themes that are addressed in the online-program are for example self-esteem, coping with relapse, establishing a structure for daily life and attention and breathing exercises as well as depression-specific topics such as negative thoughts management and arranging and maintaining social contacts. In addition, participants were able to participate in exchange with peers via an internal closed forum.
  Interventions: Behavioral: Selfapy with additional peer support
- No intervention: waitlist-control group (No Intervention): The participants of the wait-list control condition do not receive any new intervention during the intervention period of 9 weeks, but may continue any treatment that has already been started before, including medication. Participants in the wait-list control condition receive full access to the program after completion of the post-assessment.
- Online self-help program with therapeutic guidance (Experimental): The intervention group receives the login data for the online program directly following the baseline assessment. The program consists of 9 modules with many interactional exercises. Themes that are addressed in the online-program are for example self-esteem, coping with relapse, establishing a structure for daily life and attention and breathing exercises as well as depression-specific topics such as negative thoughts management and arranging and maintaining social contacts. In addition, participants were able to talk about personal experiences and difficulties concerning the program on a weekly basis with a therapeutic guide on the phone.
  Interventions: Behavioral: Selfapy with therapeutic guidance

INTERVENTIONS:
Behavioral: Selfapy with therapeutic guidance — The program consists of 9 modules with many interactional exercises. Themes that are addressed in the online-program are for example self-esteem, coping with relapse, establishing a structure for daily life and attention and breathing exercises as well as depression-specific topics such as negative thoughts management and arranging and maintaining social contacts. In addition, participants were able to talk about personal experiences with a therapeutic guide.
  Arms: Online self-help program with therapeutic guidance
Behavioral: Selfapy with additional peer support — The program consists of 9 modules with many interactional exercises. Themes that are addressed in the online-program are for example self-esteem, coping with relapse, establishing a structure for daily life and attention and breathing exercises as well as depression-specific topics such as negative thoughts management and arranging and maintaining social contacts. In addition, participants were able to participate in exchange with peers via an internal closed forum.
  Arms: Online self-help program with additional peer support

SUMMARY:
The study examines the effectiveness of a internet-based self-help-program called Selfapy for individuals who are experiencing mental stress. The main objective of the study is to investigate the extent to which Selfapy leads to a significant reduction in depressive symptoms. As this study is the first to evaluate the program Selfapy, also quality of life and acceptance of the program are evaluated. The study is conducted as a randomized-controlled trial with parallel assignment into three conditions. The groups were organized into one wait-list control group and two groups receiving access to Selfapy with different levels of guidance.

DETAILED DESCRIPTION:
The study examines the effectiveness of a internet-based self-help-program called Selfapy for individuals who are experiencing mental stress. The main objective of the study is to investigate the extent to which Selfapy leads to a significant reduction in depressive symptoms. As this study is the first to evaluate the program Selfapy, also quality of life and acceptance of the program are evaluated. The primary outcome is the PHQ-9 as a measure of the severity of depressive symptoms, combined with the BDI-II. Secondary outcomes are rates of quality of life and satisfaction with the program, which were measured with the WHOQOL-BREF and ZUF-8. The study is conducted as a randomized-controlled trial with parallel assignment into three conditions over the course of three months. The groups were organized into one wait-list control group, one that received Selfapy with additional peer support and one that received Selfapy with therapeutic guidance.The wait-list control group received access to the program after completion of the post-survey.

ELIGIBILITY:
Inclusion Criteria:

Subjective psychological distress caused by depressive symptoms, wish for treatment, access to Internet, sufficient knowledge of the German language.

Exclusion Criteria:

Acute suicidal tendencies, lifetime diagnoses of schizophrenia or bipolar disorder, presence of neurological or dementia disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
Change in depression measured with Patient Health Questionnaire 9 - Depression module (PHQ-9) | Assesses symptoms over the last two weeks; provided at baseline and post (after 3 months); change from baseline to post is being measured
  The PHQ-9 (Kroenke et al. 2001) is made up of 9 items which could be self-rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). Major depression and other depression diagnoses according to DSM-IV can be determined according to the overall score. Sum scores of 0-4 indicate none or minimal depressive symptoms, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, and 15-27 severe depressive symptoms. Its internal consistency ranges from 0.86-0.89 (Smarr and Keefer 2011).
Change in depression measured with Beck Depression Inventory (BDI-II) | Assesses symptoms over the last two weeks; provided at baseline and post (after 3 months); change from baseline to post is being measured
  The BDI-II (Beck et al., 1996) is a 21-item self-report inventory measuring the severity of depression in adolescents and adults. Each item is rated on a four-point Likert scale ranging from 0 (symptom not present) to 3 (symptom very intense). The BDI assesses psychological and physical symptoms over the last two weeks in order to quantify levels of depression. An overall score of 0-13 indicates minimal depression, a score of 14-19 indicates mild depression, a score of 20-28 moderate depression and total scores of 29-63 suggest severe depression. The internal consistency of the BDI-II ranges from 0.79-0.90 (Smarr and Keefer 2011).

SECONDARY OUTCOMES:
Change in quality of life measured with World Health Organization Quality Of Life - abbreviated version (WHOQOL-BREF) | Assesses symptoms over the last two weeks; provided at baseline and post (after 3 months); change from baseline to post is being measured
  The WHOQOL-BREF is a shorter version of the World Health Organization Quality of Life-100 (The WHOQOL Group 1998). It is composed of 26 self-report items measuring domains such as physical health, psychological health, social relationships and environment with the aim of measuring changes in quality of life over the course of treatment. Four different types of 5-point Likert scales are applied, asking "how much", "how complete", "how often", "how good" or "how satisfied" the person felt concerning the past two weeks. The WHOQOL-BREF has an internal consistency of .70 (Skevington, Lotfy, & O'Connell, 2004).
Questionnaire to measure patient satisfaction (Fragebogen zur Patientenzufriedenheit, ZUF-8) | Assesses patient satisfaction with the program at the time of assessment; provided only at post (3 months after baseline)
  The German version of the Questionnaire to measure patient satisfaction (Fragebogen zur Patientenzufriedenheit, ZUF-8; Schmidt, Lamprecht, & Wittmann, 1989) is a self-report inventory that measures client satisfaction concerning the received treatment during inpatient stays. Each item could be answered on a 4-point Likert scale ranging from 1 (totally disagree) to 4 (totally agree). The internal consistency of the ZUF-8 ranges between 0.87-0.93 (Brähler, Schumacher, & Strauß, 2002).

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Moritz, Prof., Principal Investigator — University Medical Center Hamburg-Eppendorf, Germany
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany